CLINICAL TRIAL: NCT01329328
Title: Effect of Whole-body Vibration With or Without Localized Radiofrequency on Body Composition and Subcutaneous Fat in Obese Females
Brief Title: Whole-body Vibration With or Without Localized Radiofrequency and Body Composition in Obese Female
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: Bios S.r.l. (Industry)
Responsible Party: Principal Investigator, Carlo Zancanaro, Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VIBROB
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Obesity
Keywords: whole-body vibration; radiofrequency; muscular strength; exercise; body composition
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- CONTROL (No Intervention): NO VIBRATION EXERCISE
- VIBRATION EXERCISE (Experimental): WHOLE-BODY VIBRATION EXERCISE ON A VIBRATION DEVICE (BIOPLATE RF, BIOS, MILAN, ITALY
  Interventions: Device: vibrating platform (Bioplate RF)
- VIBRATION EXERCISE PLUS RADIOFREQUENCY ADMINISTRATION (Experimental): WHOLE-BODY VIBRATION EXERCISE ON A VIBRATION DEVICE (BIOPLATE RF, BIO, MILAN, ITALY PLUS LOCAL ADMINISTRATION OF RADIOFREQUENCY
  Interventions: Device: vibrating platform (Bioplate RF)

INTERVENTIONS:
Device: vibrating platform (Bioplate RF) — whole body vibration exercise with multiple positions, with or without localized delivery of heating radiofrequency
  Other Names: Bioplate RF vibrating platform
  Arms: VIBRATION EXERCISE; VIBRATION EXERCISE PLUS RADIOFREQUENCY ADMINISTRATION

SUMMARY:
The aim of this study is to evaluate the effect of whole-body vibration in the presence or absence of localized radiofrequency on body composition in obese female subjects. Moreover, strength tests will be performed. The study hypothesis is that whole-body vibration induces positive changes in body composition i.e., reduction of fat mass and increase of lean mass with associated increase in performance. The possible additive role of radiofrequency will also be assessed.

DETAILED DESCRIPTION:
* recruitment of female obese subjects
* baseline assessment (body composition with dual energy x-ray absorptiometry (DXA) and strength tests)
* 2-mo whole body vibration training (2 sessions a week, 30 min per session) with or without local delivery of radiofrequency (two randomly selected groups)
* final assessment (body composition with DXA and strength tests)
* data collation and analysis

ELIGIBILITY:
Inclusion Criteria:

* BMI: >25
* normal locomotion
* informed consent form signed

Exclusion Criteria:

* acute illness
* endocrine pathologies or diabetes mellitus
* vascular pathology
* pacemaker
* pregnancy

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Zancanaro, MD, Principal Investigator — Universita di Verona

RESULTS

PARTICIPANT FLOW:
Groups:
- CONTROL: CONTROL GROUP NO INTERVENTION
- WHOLE-BODY VIBRATION: EXERCISE ON A VIBRATION DEVICE (BIOPLATE RF, BIOS, MILAN, ITALY
- WHOLE-BODY VIBRATION PLUS RADIOFREQUENCY: EXERCISE ON A VIBRATION DEVICE (BIOPLATE RF,BIOS, MILAN, ITALY) PLUS LOCAL ADMINISTRATION OF RADIOFREQUENCY
Period: Overall Study
Arm/Group | CONTROL | WHOLE-BODY VIBRATION | WHOLE-BODY VIBRATION PLUS RADIOFREQUENCY
Started | 15 | 17 | 18
Completed | 13 | 13 | 15
Not Completed | 2 | 4 | 3
Not completed — Withdrawal by Subject | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- VIBRATION EXERCISE: WHOLE-BODY VIBRATION EXERCISE ON A VIBRATION DEVICE (BIOPLATE RF, BIOS, MILAN, ITALY
  vibrating platform (Bioplate RF): whole body vibration exercise with multiple positions, without localized delivery of heating radiofrequency
- VIBRATION EXERCISE PLUS RADIOFREQUENCY ADMINISTRATION: WHOLE-BODY VIBRATION EXERCISE ON A VIBRATION DEVICE (BIOPLATE RF, BIO, MILAN, ITALY PLUS LOCAL ADMINISTRATION OF RADIOFREQUENCY
  vibrating platform (Bioplate RF): whole body vibration exercise with multiple positions, with localized delivery of heating radiofrequency
- Total: Total of all reporting groups
Arm/Group | CONTROL | VIBRATION EXERCISE | VIBRATION EXERCISE PLUS RADIOFREQUENCY ADMINISTRATION | Total
Number analyzed (Participants) | 15 | 17 | 18 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (5.6) | 49.0 (5.6) | 45.4 (10.4) | 46.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 18 | 50
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Body Composition
Description: Evidence of changes in body composition (three-compartment model as assessed by dual-energy X-ray absorptiometry) after two months of whole-body vibration with or without application of localized radiofrequency
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: PECENTAGE OF WHOLE-BODY FAT
Arm/Group | CONTROL | VIBRATION EXERCISE | VIBRATION EXERCISE PLUS RADIOFREQUENCY ADMINISTRATION
Number analyzed (Participants) | 13 | 13 | 15
PECENTAGE OF WHOLE-BODY FAT | 44.8 (3.9) | 43.4 (4.1) | 44.0 (3.7)

2. Secondary Outcome: Muscular Strength
Description: evidence of changes in lower limbs muscular strength following 2 months of whole-body vibration
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: KILOGRAMS
Arm/Group | CONTROL | VIBRATION EXERCISE | VIBRATION EXERCISE PLUS RADIOFREQUENCY ADMINISTRATION
Number analyzed (Participants) | 13 | 13 | 15
KILOGRAMS | 212.0 (43.10) | 217.3 (49.9) | 213.8 (56.5)

ADVERSE EVENTS:
Time Frame: 3 MONTHS
Arm/Group | CONTROL | VIBRATION EXERCISE | VIBRATION EXERCISE PLUS RADIOFREQUENCY ADMINISTRATION
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes